CLINICAL TRIAL: NCT06564298
Title: Sintilimab Combined With Ramucirumab and Chemotherapy as First-line Treatment in Patients With Advanced Gastric Cancer With Liver Metastasis (RAMSINT): A Phase II, Single-center, Prospective Clinical Study
Brief Title: A Study on the Combination of Sintilimab, Ramucirumab and Chemotherapy for First-line Treatment of Gastric Cancer With Liver Metastasis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-654
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; Ramucirumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+Ramucirumab+SOX/XELOX (Experimental)
  Interventions: Drug: Sintilimab; Drug: Ramucirumab; Drug: SOX/XELOX

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg iv.gtt d1, every 21 days
Drug: Ramucirumab — Ramucirumab 10mg/kg iv.gtt d1, every 21 days
Drug: SOX/XELOX — SOX: Oxaliplatin 130mg/m2 iv.gtt d1, every 21 days and S-1 40mg/m2 po bid d1-14, every 21 days XELOX: Oxaliplatin 130mg/m2 iv.gtt d1, every 21 days and Capecitabine 1000mg/m2 po bid d1-14, every 21 days

SUMMARY:
The goal of this clinical trial is to observe the efficacy and safety of Sintilimab (a PD-1 inhibitor) combined with Ramucirumab (a VEGFR-2 antagonist) and chemotherapy as a first-line treatment for patients with advanced gastric cancer with liver metastasis.

* Can the combination of Sintilimab, Ramucirumab, and chemotherapy improve the prognosis of patients with AGC and liver metastases?
* What are the adverse events (AEs) associated with the use of the combination regimen of Sintilimab, Ramucirumab, and chemotherapy in patients with AGC and liver metastases?

Participants will:

* Receive a combined treatment regimen of Sintilimab, Ramucirumab, and chemotherapy (SOX (oxaliplatin and S-1) or XELOX (oxaliplatin and capecitabine)), administered every 21 days for up to 6 cycles. Following the completion of 6 cycles, maintenance therapy with Sintilimab and oral chemotherapy agents (capecitabine or S-1) with or without Ramucirumab will be administered until disease progression.
* Imaging assessments will be performed at baseline, after every 2 cycles of treatment, and every 3 months following the completion of 6 cycles of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical study; full understanding and informed consent to this study by signing the Informed Consent Form (ICF); willingness to follow and ability to complete all trial procedures.
2. Patients with histologically or cytologically confirmed, unresectable, or who refuse surgical resection of locally advanced, recurrent, or metastatic gastric and gastroesophageal junction (GEJ) adenocarcinoma (including signet-ring cell carcinoma, mucinous adenocarcinoma, hepatoid adenocarcinoma, etc.). (Note: For patients who relapse after neoadjuvant/adjuvant therapy, the time from the end of neoadjuvant/adjuvant therapy to disease relapse must be more than 6 months.)
3. Patients, except those with recurrent disease after neoadjuvant/adjuvant therapy, must not have previously received systemic treatment.
4. Participants must be histologically confirmed as having HER2-negative gastric cancer, GEJ cancer, or esophageal adenocarcinoma.
5. There must be at least one measurable lesion in the liver assessed by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) that can undergo repeat radiological evaluation; the radiological tumor assessment should be performed within 28 days prior to randomization.
6. The Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2 within 7 days prior to the first dose of medication.
7. Availability of representative tumor tissue specimens, blood samples, and fecal samples for exploratory research.
8. Main organ functions must be normal, meeting the following criteria:

Liver Function Alanine Aminotransferase (ALT) ≤5.0 × ULN Aspartate Aminotransferase (AST) ≤5.0 × ULN

Exclusion Criteria:

1. History of other active malignancies within the past 5 years or currently having other active malignancies. Treated localized tumors, such as basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, and breast carcinoma in situ, are eligible for inclusion.
2. Underwent surgery within 4 weeks prior to the start of the study treatment.
3. Known history of severe allergy to any monoclonal antibodies or excipients.
4. Previous use of PD-1 inhibitors, LAG-3 inhibitors, CTLA-4 inhibitors, or any other antibodies or drug treatments targeting T-cell co-stimulation or immune checkpoint pathways, including previous receipt of anti-tumor vaccines or other immunostimulatory anti-tumor therapies.
5. Previous exposure to VEGF (vascular endothelial growth factor) or VEGFR inhibitors or any anti-angiogenesis medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 12 months
  ORR was defined as the proportion of participants whose tumor volume decreases to a predefined value and can maintain the minimum duration requirements, which is the sum of the rates of Complete Response (CR) and Partial Response (PR) according to RECIST 1.1 based on investigator assessment.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 12 months
  DCR was defined as the percentage of the participants who achieve either a response (PR + CR) or Stable Disease (SD) after treatment and can maintain the minimum duration requirements according to RECIST 1.1 based on investigator assessment.
Progression-free Survival (PFS) | Up to approximately 16 months
  PFS was defined as the time from the start of treatment to disease progression according to RECIST 1.1 based on investigator assessment, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 16 months
  OS was defined as the time from enrollment to death due to any cause.
Incidence of adverse events and serious adverse events (AEs) | Up to approximately 16 months
  Categorized according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE 5.0). Descriptive statistical analysis is primarily used to list and describe the AEs that occurred during this trial.